CLINICAL TRIAL: NCT03854071
Title: Development of Novel Physiological CMR Methods in Health and Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STH20184
Record Dates: First submitted 2019-02-19; First posted 2019-02-26 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure; Pulmonary Hypertension; Myocardial Infarction; Coronary Artery Disease
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary; Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients will be selected in each group by the clinical specialist/research team as per the published guidelines and local protocols - Group 1, Group 2, Group 3, Group 4 and Group 5.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Other): Heart failure patients with preserved ejection fraction
  Interventions: Other: intravenous fluid challenge
- Group 2 (Other): Heart failure patients with reserved ejection fraction
  Interventions: Other: intravenous fluid challenge
- Group 3 (Other): Patients with pulmonary hypertension
  Interventions: Other: intravenous fluid challenge
- Group 4 (Other): Patients with acute myocardial infarction
  Interventions: Other: intravenous fluid challenge
- Group 5 (Other): Patients with suspected but not treated coronary artery disease
  Interventions: Other: intravenous fluid challenge
- Group 6 (Other): Healthy Volunteers
  Interventions: Other: intravenous fluid challenge

INTERVENTIONS:
Other: intravenous fluid challenge — Patients will undergo a receive a pre-load increasing stress test with intravenous fluids depending on tolerability

SUMMARY:
Physiological cardiovascular stress test plays a crucial role in the assessment of patients with suspected heart disease. There are several methods of cardiac physiological stress tests and each of them offer varied insight into cardiac physiological adaptation: passive leg raise, intra-venous fluid challenge, pharmacological stressors and physical exercise stress test. Echocardiography, which is the mainstay for the non-invasive rest/stress assessment of the left ventricular (LV) haemodynamics has several limitations. Novel methods of CMR imaging allow to map intra-cardiac flow in three-dimension using novel flow acquisitions. These novel flow acquisitions are called four-dimensional flow CMR, where the fourth dimension is time. Additionally, traditional cine CMR imaging for functional assessment can now be done without breath-holds using advanced acceleration methods, allowing them to be used during exercise. A comprehensive understanding of functional-flow coupling at rest, during increased pre-load (fluid challenge) to the heart or during exercise, is lacking in the literature. There is an important need to validate these novel CMR methods for developing mechanistic insight into physiological cardiac adaptation to increased pre-load or to exercise in health and how it alters in heart disease.

DETAILED DESCRIPTION:
For this study, the investigators will perform comprehensive physiological CMR in healthy volunteers and patients with suspected or known heart disease (coronary artery disease and heart failure). A sub-set of patients will have follow-up scans after they receive treatment to investigate the therapeutic target role of these physiological CMR metrics.

Patients who have given informed consent for this research will receive one physiological stress test depending on the clinical context. There will be 5 clinical subgroups to which patients will be recruited to:

Group 1. Heart failure with preserved ejection fraction (HFpEF), Group 2. Heart failure with reserved ejection fraction (HFrEF), Group 3. Pulmonary hypertension (PH), Group 4. Acute myocardial infarction (AMI) and Group 5. Suspected but not treated coronary artery disease (sCAD).

Patients will be selected in each group by the clinical specialist/research team as per the published guidelines and local protocols - Group 1 and 2 (19), Group 3 (20), Group 4 (21) and Group 5 (22).

First 4 groups of patients will receive pre-load increasing stress test (either passive leg raise or equivalent 500mls intravenous fluid challenge depending on the tolerability). This will be done to investigate if increase in pre-load will help unravel subtle dysfunction which is not apparent at euvolemic state. AMI patients may also receive ischaemia testing stress CMR depending on the main clinically question needed to answer. Patients with sCAD will receive clinically relevant pharmacological stress test (dobutamine, adenosine or regadenoson, inhaled nitric oxide) to diagnose ischaemia.

Healthy volunteers who have given informed consent will receive matched physiological stress test so that head-on comparison can be made with the relevant patient cohort. The CMR scan protocol will involve minimal breath-holds and will be patient-friendly. This is achieved by using accelerated, advanced cine and late gadolinium enhancement (LGE)-imaging techniques which require fewer breath-holds and shorter scan. All CMR stress studies will be supervised by an Advanced Life Support (ALS) certified doctor.

The CMR protocol for healthy volunteers will include the following components (45 minutes):

1. Survey
2. Baseline cine imaging for functional imaging (rest)
3. Tissue characterisation with native T1-mapping (rest)
4. 4D flow CMR (rest)
5. Record blood pressure, heart rate and oxygen saturation
6. Start of physiological stress (increase pre-load or pharmacological stressors)
7. 4D flow CMR (stress, at low-moderate intensity exercise aiming for heart rate up to 110bpm only)
8. Functional cines (stress, at low-moderate intensity exercise aiming for heart rate up to 110bpm only)
9. Record blood pressure, heart rate and oxygen saturation
10. First pass perfusion imaging (only if adenosine/regadenoson used for myocardial hyperaemia)
11. Record blood pressure, heart rate and oxygen saturation
12. Gadolinium contrast injection
13. Early/Late gadolinium enhancement imaging in short-axis
14. Post contrast T1-mapping End of study

For patient's receiving clinical CMR scans, the 'bolt-on' stress CMR protocol will include the following components (20-25minutes):

1. 4D flow CMR (rest)
2. Record blood pressure, heart rate and oxygen saturation
3. Start of physiological stress (increase pre-load or pharmacological stressors)
4. 4D flow CMR (stress, at low-moderate intensity exercise aiming for heart rate up to 110bpm only)
5. Functional cines (stress, at low-moderate intensity exercise aiming for heart rate up to 110bpm only)
6. Record blood pressure, heart rate and oxygen saturation
7. First pass perfusion imaging (only if adenosine/regadenoson used for myocardial hyperaemia)
8. Record blood pressure, heart rate and oxygen saturation

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers age 20 to 80, recruited from Sheffield Teaching Hospitals staff members
* Patients age 20 to 80 with suspected or known heart disease (group 1 to 5)
* Capable of giving written informed consent

Exclusion Criteria:

* Inability to perform the study protocol secondary to severe heart failure requiring IV therapy
* Patients recruited in the suspected CAD and acute myocardial infarction arms of the study and in need for detection of ischaemia should not have any past medical history of MI, ACS or cardiomyopathy
* Patients with significant valvular heart disease will be excluded from any patient group
* Patient with in atrial fibrillation will be excluded
* Contraindication to MRI (as per standard MRI screening questionnaire issued to patients prior to clinical MRI procedures)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
4D CMR Flow | Through study completion, average 5 years
  The primary outcome measures will include 4D flow CMR derived mitral inflow diastolic parameter: E/A ratio. This parameter will be quantified once both at rest and during physiological stress.

SECONDARY OUTCOMES:
Secondary 4D CMR Flow | Through study completion, average 5 years
  Other 4D flow CMR derived outcome metrics will include mitral, tricuspid and pulmonary valve flow quantification - net forward flow (mls), E-velocity (cm/sec), E-velocity deceleration time (msec, both for mitral and tricuspid), A-velocity (cm/sec) and valvular regurgitation (mls).
Volumetric and functional parameters | Through study completion, average 5 years
  2) Right and left heart volumetric and functional parameters: end-diastolic and end-systolic volumes; ejection fraction

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS FT, Sheffield, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Obokata M, Kane GC, Reddy YN, Olson TP, Melenovsky V, Borlaug BA. Role of Diastolic Stress Testing in the Evaluation for Heart Failure With Preserved Ejection Fraction: A Simultaneous Invasive-Echocardiographic Study. Circulation. 2017 Feb 28;135(9):825-838. doi: 10.1161/CIRCULATIONAHA.116.024822. Epub 2016 Dec 30. PMID 28039229
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Popescu BA, Waggoner AD. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2016 Apr;29(4):277-314. doi: 10.1016/j.echo.2016.01.011. No abstract available. PMID 27037982
- [Background] Sharifov OF, Schiros CG, Aban I, Denney TS, Gupta H. Diagnostic Accuracy of Tissue Doppler Index E/e' for Evaluating Left Ventricular Filling Pressure and Diastolic Dysfunction/Heart Failure With Preserved Ejection Fraction: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2016 Jan 25;5(1):e002530. doi: 10.1161/JAHA.115.002530. PMID 26811160
- [Background] Franke A. The stress echo dilemma: time counts, but image quality too. Eur Heart J. 2006 Jul;27(14):1646-7. doi: 10.1093/eurheartj/ehl091. Epub 2006 Jun 16. No abstract available. PMID 16782718
- [Background] Westenberg JJ, Roes SD, Ajmone Marsan N, Binnendijk NM, Doornbos J, Bax JJ, Reiber JH, de Roos A, van der Geest RJ. Mitral valve and tricuspid valve blood flow: accurate quantification with 3D velocity-encoded MR imaging with retrospective valve tracking. Radiology. 2008 Dec;249(3):792-800. doi: 10.1148/radiol.2492080146. Epub 2008 Oct 10. PMID 18849503
- [Background] Crandon S, Elbaz MSM, Westenberg JJM, van der Geest RJ, Plein S, Garg P. Clinical applications of intra-cardiac four-dimensional flow cardiovascular magnetic resonance: A systematic review. Int J Cardiol. 2017 Dec 15;249:486-493. doi: 10.1016/j.ijcard.2017.07.023. Epub 2017 Sep 28. PMID 28964555
- [Background] Pedrizzetti G, La Canna G, Alfieri O, Tonti G. The vortex--an early predictor of cardiovascular outcome? Nat Rev Cardiol. 2014 Sep;11(9):545-53. doi: 10.1038/nrcardio.2014.75. Epub 2014 Jun 3. PMID 24889521
- [Background] Carlsson M, Toger J, Kanski M, Bloch KM, Stahlberg F, Heiberg E, Arheden H. Quantification and visualization of cardiovascular 4D velocity mapping accelerated with parallel imaging or k-t BLAST: head to head comparison and validation at 1.5 T and 3 T. J Cardiovasc Magn Reson. 2011 Oct 4;13(1):55. doi: 10.1186/1532-429X-13-55. PMID 21970399
- [Background] Eriksson J, Bolger AF, Ebbers T, Carlhall CJ. Four-dimensional blood flow-specific markers of LV dysfunction in dilated cardiomyopathy. Eur Heart J Cardiovasc Imaging. 2013 May;14(5):417-24. doi: 10.1093/ehjci/jes159. Epub 2012 Aug 8. PMID 22879457
- [Background] Eriksson J, Dyverfeldt P, Engvall J, Bolger AF, Ebbers T, Carlhall CJ. Quantification of presystolic blood flow organization and energetics in the human left ventricle. Am J Physiol Heart Circ Physiol. 2011 Jun;300(6):H2135-41. doi: 10.1152/ajpheart.00993.2010. Epub 2011 Mar 18. PMID 21421820
- [Background] Watanabe H, Sugiura S, Hisada T. The looped heart does not save energy by maintaining the momentum of blood flowing in the ventricle. Am J Physiol Heart Circ Physiol. 2008 May;294(5):H2191-6. doi: 10.1152/ajpheart.00041.2008. Epub 2008 Mar 7. PMID 18326797
- [Background] Kanski M, Arvidsson PM, Toger J, Borgquist R, Heiberg E, Carlsson M, Arheden H. Left ventricular fluid kinetic energy time curves in heart failure from cardiovascular magnetic resonance 4D flow data. J Cardiovasc Magn Reson. 2015 Dec 20;17:111. doi: 10.1186/s12968-015-0211-4. PMID 26685664
- [Background] Wong J, Chabiniok R, deVecchi A, Dedieu N, Sammut E, Schaeffter T, Razavi R. Age-related changes in intraventricular kinetic energy: a physiological or pathological adaptation? Am J Physiol Heart Circ Physiol. 2016 Mar 15;310(6):H747-55. doi: 10.1152/ajpheart.00075.2015. Epub 2016 Jan 8. PMID 26747496
- [Background] Ie EH, Vletter WB, ten Cate FJ, Nette RW, Weimar W, Roelandt JR, Zietse R. Preload dependence of new Doppler techniques limits their utility for left ventricular diastolic function assessment in hemodialysis patients. J Am Soc Nephrol. 2003 Jul;14(7):1858-62. doi: 10.1097/01.asn.0000072745.94551.fc. PMID 12819246
- [Background] Zhou BY, Xie MX, Wang J, Wang XF, Lv Q, Liu MW, Kong SS, Zhang PY, Liu JF. Relationship between the abnormal diastolic vortex structure and impaired left ventricle filling in patients with hyperthyroidism. Medicine (Baltimore). 2017 Apr;96(17):e6711. doi: 10.1097/MD.0000000000006711. PMID 28445281
- [Background] Kheradvar A, Assadi R, Falahatpisheh A, Sengupta PP. Assessment of transmitral vortex formation in patients with diastolic dysfunction. J Am Soc Echocardiogr. 2012 Feb;25(2):220-7. doi: 10.1016/j.echo.2011.10.003. Epub 2011 Nov 17. PMID 22099070
- [Background] van der Geest RJ, Garg P. Advanced Analysis Techniques for Intra-cardiac Flow Evaluation from 4D Flow MRI. Curr Radiol Rep. 2016;4:38. doi: 10.1007/s40134-016-0167-7. Epub 2016 May 20. PMID 27390626
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M; ESC Scientific Document Group. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Heart J. 2016 Jan 1;37(1):67-119. doi: 10.1093/eurheartj/ehv317. Epub 2015 Aug 29. No abstract available. PMID 26320113
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for Universal Definition of Myocardial Infarction; Authors/Task Force Members Chairpersons; Thygesen K, Alpert JS, White HD; Biomarker Subcommittee; Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA; ECG Subcommittee; Chaitman BR, Clemmensen PM, Johanson P, Hod H; Imaging Subcommittee; Underwood R, Bax JJ, Bonow JJ, Pinto F, Gibbons RJ; Classification Subcommittee; Fox KA, Atar D, Newby LK, Galvani M, Hamm CW; Intervention Subcommittee; Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J; Trials & Registries Subcommittee; Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML; Trials & Registries Subcommittee; Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G; Trials & Registries Subcommittee; Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D; Trials & Registries Subcommittee; Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG); Bax JJ, Baumgartner H, Ceconi C, Dean V, Deaton C, Fagard R, Funck-Brentano C, Hasdai D, Hoes A, Kirchhof P, Knuuti J, Kolh P, McDonagh T, Moulin C, Popescu BA, Reiner Z, Sechtem U, Sirnes PA, Tendera M, Torbicki A, Vahanian A, Windecker S; Document Reviewers; Morais J, Aguiar C, Almahmeed W, Arnar DO, Barili F, Bloch KD, Bolger AF, Botker HE, Bozkurt B, Bugiardini R, Cannon C, de Lemos J, Eberli FR, Escobar E, Hlatky M, James S, Kern KB, Moliterno DJ, Mueller C, Neskovic AN, Pieske BM, Schulman SP, Storey RF, Taubert KA, Vranckx P, Wagner DR. Third universal definition of myocardial infarction. J Am Coll Cardiol. 2012 Oct 16;60(16):1581-98. doi: 10.1016/j.jacc.2012.08.001. Epub 2012 Sep 5. No abstract available. PMID 22958960
- [Background] Task Force Members; Montalescot G, Sechtem U, Achenbach S, Andreotti F, Arden C, Budaj A, Bugiardini R, Crea F, Cuisset T, Di Mario C, Ferreira JR, Gersh BJ, Gitt AK, Hulot JS, Marx N, Opie LH, Pfisterer M, Prescott E, Ruschitzka F, Sabate M, Senior R, Taggart DP, van der Wall EE, Vrints CJ; ESC Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Knuuti J, Valgimigli M, Bueno H, Claeys MJ, Donner-Banzhoff N, Erol C, Frank H, Funck-Brentano C, Gaemperli O, Gonzalez-Juanatey JR, Hamilos M, Hasdai D, Husted S, James SK, Kervinen K, Kolh P, Kristensen SD, Lancellotti P, Maggioni AP, Piepoli MF, Pries AR, Romeo F, Ryden L, Simoons ML, Sirnes PA, Steg PG, Timmis A, Wijns W, Windecker S, Yildirir A, Zamorano JL. 2013 ESC guidelines on the management of stable coronary artery disease: the Task Force on the management of stable coronary artery disease of the European Society of Cardiology. Eur Heart J. 2013 Oct;34(38):2949-3003. doi: 10.1093/eurheartj/eht296. Epub 2013 Aug 30. No abstract available. PMID 23996286
- [Background] Monmeneu Menadas JV, Lopez-Lereu MP, Estornell Erill J, Garcia Gonzalez P, Igual Munoz B, Maceira Gonzalez A. Pharmacological stress cardiovascular magnetic resonance: feasibility and safety in a large multicentre prospective registry. Eur Heart J Cardiovasc Imaging. 2016 Mar;17(3):308-15. doi: 10.1093/ehjci/jev153. Epub 2015 Jun 23. PMID 26108417
- [Background] Mertes H, Sawada SG, Ryan T, Segar DS, Kovacs R, Foltz J, Feigenbaum H. Symptoms, adverse effects, and complications associated with dobutamine stress echocardiography. Experience in 1118 patients. Circulation. 1993 Jul;88(1):15-9. doi: 10.1161/01.cir.88.1.15. PMID 8319327
- [Background] Garg P, Westenberg JJM, van den Boogaard PJ, Swoboda PP, Aziz R, Foley JRJ, Fent GJ, Tyl FGJ, Coratella L, ElBaz MSM, van der Geest RJ, Higgins DM, Greenwood JP, Plein S. Comparison of fast acquisition strategies in whole-heart four-dimensional flow cardiac MR: Two-center, 1.5 Tesla, phantom and in vivo validation study. J Magn Reson Imaging. 2018 Jan;47(1):272-281. doi: 10.1002/jmri.25746. Epub 2017 May 4. PMID 28470915